CLINICAL TRIAL: NCT01009840
Title: A Phase 2a Study of Once Daily Intravenous Busulfan With Bortezomib, Followed by an Autologous Hematopoietic Stem Cell Transplant (HSCT) in Subjects With Relapsed Multiple Myeloma After Prior Autologous HSCT
Brief Title: IV Busulfan Plus Bortezomib Conditioning Regimen for Second Autologous Stem Cell Transplant in Multiple Myeloma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 273-08-205
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Results first posted 2014-08-07 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Bone marrow transplant; Stem cell transplant; Busulfan; Bortezomib
MeSH Terms: conditions — Multiple Myeloma | interventions — Busulfan; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IV busulfan (Experimental): Intravenous (IV) busulfan was administered as a single daily 3-hour continuous infusion based on the PK-directed dose recommendation for 4 days beginning on Day -5 followed by a single bortezomib 1.3 mg/m^2 dose administered as a 3 to 5-second bolus IV injection on Day -1 prior to HSCT.
  Interventions: Drug: IV busulfan; Drug: bortezomib; Procedure: Autologous Hematopoietic Stem Cell Transplant (HSCT)

INTERVENTIONS:
Drug: IV busulfan — PK-directed dosing of IV busulfan for 4 days
  Other Names: Busulfex®
Drug: bortezomib — Single IV bortezomib at a dose of 1.3 mg/m^2.
  Other Names: Velcade®
Procedure: Autologous Hematopoietic Stem Cell Transplant (HSCT)

SUMMARY:
Study for the outcome and safety of individualized busulfan dosing with bortezomib for patients preparing for a second stem cell transplant to treat multiple myeloma.

DETAILED DESCRIPTION:
Evaluation of six-month response in relapsed multiple myeloma subjects, who have had a prior autologous HSCT (greater than one year previously) receiving an IV busulfan-based conditioning regimen with the combination of pharmacokinetic (PK)-guided IV busulfan dosing and bortezomib, followed by a second autologous HSCT.

Assessment of the safety profile of this conditioning regimen will also be completed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years, inclusive.
2. Subjects must have multiple myeloma which requires treatment for relapsed disease and are eligible for the planned autologous HSCT.
3. Subjects must have had one previous autologous HSCT, at least one year prior to the planned autologous HSCT in this study.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
5. Negative beta-human chorionic gonadotropin (β-HCG) pregnancy test in all women of child-bearing potential.
6. Subjects who are surgically sterile (ie, have undergone orchidectomy or hysterectomy); female subjects who have been postmenopausal for at least 12 consecutive months; or subjects who agree to remain abstinent or to practice double-barrier forms of birth control from trial screening through 30 days (for females) and 90 days (for males) from the last dose of the investigational medicinal product (IMP). If employing birth control, two of the following precautions must be used: vasectomy, tubal ligation, vaginal diaphragm, intrauterine device (IUD), birth control pill, birth control implant, condom, or sponge with spermicide.
7. Subjects in whom the minimum stem cell dose of 2.0 x 10^6 cluster of differentiation 34 (CD34)+ cells/kg has been collected.
8. Ability to provide written informed consent prior to initiation of any study-related procedures, and ability, in the opinion of the Principal Investigator, to comply with all requirements of the study.

Exclusion Criteria:

1. Prior treatment history of allogeneic HSCT for any medical reason, not limited to myeloma treatment.
2. Prior treatment history of more than one autologous HSCT or high-dose chemotherapy with stem cell rescue for any medical reason, not limited to myeloma treatment.
3. Prior treatment with busulfan or gemtuzumab ozogamicin for any reason.
4. Presence of a t(4;14) or p53 gene deletion as determined by fluorescence in situ hybridization (FISH) during the screening process or documented t(4; 14) or p53 gene deletion obtained during a time of active disease by any method.
5. Systemic amyloidosis.
6. Known allergy to boron or any components of bortezomib.
7. Left ventricular ejection fraction (LVEF) < 45% as measured by either multi-gated acquisition scan (MUGA) or echocardiogram (ECHO) performed within 75 days prior to day of busulfan test dose. If cyclophosphamide was used for stem cell harvest, an ECHO or MUGA must be done prior to enrollment to confirm adequate cardiac function.
8. Uncontrolled arrhythmia or symptomatic cardiac disease at the time of screening.
9. Symptomatic pulmonary disease, based on Forced Expiratory Volume in 1 Second (FEV1), Forced Vital Capacity (FVC) or Diffusing Capacity of the Lung for Carbon Monoxide (DLCO) < 50% of predicted (corrected for hemoglobin) measured within 75 days prior to day of busulfan test dose.
10. Aspartate transaminase (AST)/alanine transaminase (ALT) ≥ 3 x the upper limit of normal (ULN),
11. History of elevated total serum bilirubin >2 mg/dL that had been caused by previous chemotherapy at any point, or total bilirubin > 2.0 mg/dL at the time of screening with the exception of Gilbert's disease.
12. Hepatic synthetic dysfunction evident International Normalized Ratio (INR) ≥ 2.0 at the time of screening.
13. Any previous history of fulminant liver failure, cirrhosis, alcoholic hepatitis, esophageal varices, hepatic encephalopathy, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, and symptomatic biliary disease.
14. Prior total body irradiation therapy or radiation therapy directly applied to the liver.
15. Known history of or current hepatitis B, hepatitis C, HIV, or uncontrolled active infection of any kind at the time of test dose. If serology antibody studies are positive, a quantitative polymerase chain reaction (PCR) must be completed to confirm lack of active infection.
16. Serum creatinine >2.0 mg/dL at the time of Screening.
17. ≥ Grade 1 neuropathy with pain, or > Grade 2 neuropathy without pain (subjects with neuropathy caused by a previous regimen that is recovered to ≤ Grade 2 and stable without pain may be included).
18. Women who are pregnant or lactating.
19. Current or history of drug and/or alcohol abuse.
20. Use of other investigational therapies within 30 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (11):
  - Arizona Cancer Center, Tucson, Arizona
  - Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Maryland School of Medicine - Marlene & Stewart Greenebaum Cancer Center, Baltimore, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Pennsylvania -Abramson Cancer Center, Philadelphia, Pennsylvania
  - The Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - South Texas Veterans Health Care System, San Antonio, Texas
  - Texas Transplant Physician Group, PLLC, San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
- Canada (2):
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Princess Margaret Hospital, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Groups:
- IV Busulfan: Intravenous (IV) busulfan was administered as a single daily 3-hour continuous infusion based on the pharmacokinetic (PK)-directed dose recommendation for 4 days beginning on Day -5 followed by a single bortezomib 1.3 mg/m^2 dose administered as a 3 to 5-second bolus IV injection on Day -1 prior to hematopoietic stem cell transplant (HSCT).
Period: Overall Study
Arm/Group | IV Busulfan
Started | 30
Completed | 16
Not Completed | 14
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 4
Not completed — Subject Met Withdrawal Criteria | 7
Not completed — Subject was Withdrawn by Investigator | 1
Not completed — Subject Withdrew Consent to Participate | 1

BASELINE CHARACTERISTICS:
Arm/Group | IV Busulfan
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Disease Response at Month 6
Description: The percentage of participants reported in each disease category by International Myeloma Working Group (IMWG) uniform response criteria for Multiple Myeloma 6 months after autologous Hematopoietic stem cell transplant. Overall Disease Response categories were: [stringent Complete Response (sCR)=CR + normal Free Light Chain (FLC) ratio + absence of clonal cells in bone marrow], [Complete Response (CR)=Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and ≤5% plasma cells in bone marrow], [Very Good Partial Response (VGPR)=Serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein + urine M-protein level <100 mg/24 hour], [Partial Response (PR)=≥50% reduction of serum M-protein and reduction in 24 hour urine M-protein by ≥90% or to <200 mg per 24 hour], [Stable Disease (SD)=Not meeting criteria for CR, VGPR, PR or progressive disease] or [Progressive Disease (PD)].
Time Frame: 6 Months
Population: Intent-to-treat population included all participants who received the PK-directed IV busulfan followed by autologous HSCT.
Measure: Number; unit: Percentage of participants
Arm/Group | IV Busulfan
Number analyzed (Participants) | 30
Percentage of participants
  sCR or CR or VGPR | 20.0
  PR or SD or PD | 70.0
  Not Assessed | 10.0

2. Secondary Outcome: Overall Survival
Description: Overall Survival was defined as the time in days from transplantation to death due to all causes.
Time Frame: 6 Months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | IV Busulfan
Number analyzed (Participants) | 30
Days | NA [NA to NA] — Median overall survival could not be estimated as follow-up was restricted to 6 months post transplant.

3. Secondary Outcome: Percentage of Participants With Overall Survival Events
Description: Overall Survival Event was death.
Time Frame: 6 Months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | IV Busulfan
Number analyzed (Participants) | 30
Percentage of participants | 13.3

4. Secondary Outcome: Progression-free Survival
Description: Progression-free Survival (PFS) defined as the time from transplantation to the occurrence of the event that was death or first recurrence of progressive disease (PD) by IMWG criteria. PD was defined as an Increase of ≥25% from the lowest response value in any one or more of the following: 1)Serum M-component and/or (the absolute increase must be ≥0.5 g/dL), 2)Urine M-component and/or (the absolute increase must be ≥200 mg/24 hr), 3)In patients without measurable serum and urine M-protein levels; the difference between involved and uninvolved FLC levels. The absolute increase must be >10 mg/dL, 4)Bone marrow plasma cell percentage; the absolute percentage must be ≥10%, 5)Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas and/or 6)Development of hypercalcaemia that can be attributed solely to the plasma cell proliferative diso
Time Frame: 6 Months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | IV Busulfan
Number analyzed (Participants) | 30
Days | 191 [92 to NA] — The upper limit of the 95% CI could not be estimated. Follow-up was restricted to 6 months post transplant.

5. Secondary Outcome: Percentage of Participants With Progression-free Survival Events
Description: Progression-free survival events are death or first recurrence of progressive disease by International Myeloma Working Group Criteria.
Time Frame: 6 Months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | IV Busulfan
Number analyzed (Participants) | 30
Percentage of participants | 50.0

6. Secondary Outcome: Percent Change in IV Busulfan Dose
Description: The percent change in dose is relative to the busulfan dose administered at the Baseline Visit (Day -12 to -9) when a dose of 0.8 mg/kg was administered and on Day -5 when the Seattle Cancer Care Alliance recommended PK-adjusted dose was administered.
Time Frame: Baseline (Day -12 to -9), Day -5
Population: as for outcome 1
Measure: Median (Full Range); unit: Percent change
Arm/Group | IV Busulfan
Number analyzed (Participants) | 30
Percent change | 7.55 [-26.00 to 47.50]

7. Secondary Outcome: Ratio Area Under Curve (AUC)/Target AUC
Description: A test dose of IV busulfan 0.8 mg/kg was infused at Baseline (Day -12 to -9) to verify a target busulfan integrated AUC of 20,000 μM*min with a range of 16,000 to 24,000. If necessary the dose could be adjusted. The PK-directed dose recommendation based on the test dose was administered at Day -5. Blood samples for PK analysis were collected at 0, 15, 30 minutes after the End of Infusion and 240, 300, 360 minutes after start of the infusion. Gas chromatography with mass selective detection (GC-MS) was used to determine the busulfan level in plasma. The ratio was calculated: AUC/Target AUC.
Time Frame: Baseline (Day -12 to -9), Day -5
Population: as for outcome 1
Measure: Median (Full Range); unit: Ratio
Arm/Group | IV Busulfan
Number analyzed (Participants) | 30
Ratio | 1.00 [0.89 to 1.19]

8. Secondary Outcome: Percent Difference Between Area Under Curve (AUC) and Target AUC
Description: A test dose of IV busulfan 0.8 mg/kg was infused at Baseline (Day -12 to -9) to verify a target busulfan integrated AUC of 20,000 μM*min with a range of 16,000 to 24,000. If necessary the dose could be adjusted. The PK-directed dose recommendation based on the test dose was administered at Day -5. Blood samples for PK analysis were collected at 0, 15, 30 minutes after the End of Infusion and 240, 300, 360 minutes after start of the infusion. GC-MS was used to determine the busulfan level in plasma. The percent difference was calculated between AUC and the Target AUC.
Time Frame: Baseline (Day -12 to -9), Day -5
Population: as for outcome 1
Measure: Median (Full Range); unit: Percent difference
Arm/Group | IV Busulfan
Number analyzed (Participants) | 30
Percent difference | -0.22 [-10.97 to 18.55]

9. Secondary Outcome: Percentage of Participants With Transplant-Related Mortality
Description: The percentage of participants with death related to transplant.
Time Frame: 6 Months
Population: Safety population included all participants who received IV busulfan.
Measure: Number; unit: Percentage of participants
Arm/Group | IV Busulfan
Number analyzed (Participants) | 30
Percentage of participants | 3.3

10. Secondary Outcome: Percentage of Participants With Hepatic Veno-Occlusive Disease Based on Baltimore Criteria
Description: The Baltimore criteria for veno-occlusive disease was defined as the development of hyperbilirubinemia with serum bilirubin > 2 mg/dl within 21 days after transplantation and at least 2 of the following clinical signs and symptoms: (1) hepatomegaly, usually painful, (2) > 5% weight gain, or (3) ascites.
Time Frame: 6 Months
Population: Safety population included all participants who received IV busulfan.
Measure: Number; unit: Percentage of participants
Arm/Group | IV Busulfan
Number analyzed (Participants) | 30
Percentage of participants | 0.0

ADVERSE EVENTS:
Arm/Group | IV Busulfan
Serious Adverse Events (participants affected / at risk) | 18/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IV Busulfan (N=30)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 2
Multi-organ failure (General disorders) | 1
Pyrexia (General disorders) | 3
Bacterial sepsis (Infections and infestations) | 1
Bronchitis bacterial (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Tinea versicolour (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Cranial neuropathy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Venoocclusive disease (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IV Busulfan (N=30)
Anaemia (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 17
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Palpitations (Cardiac disorders) | 4
Sinus tachycardia (Cardiac disorders) | 2
Tachycardia (Cardiac disorders) | 5
Dry eye (Eye disorders) | 2
Vision blurred (Eye disorders) | 3
Abdominal discomfort (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 4
Anal inflammation (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 13
Diarrhoea (Gastrointestinal disorders) | 26
Dry mouth (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 6
Flatulence (Gastrointestinal disorders) | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3
Hematochezia (Gastrointestinal disorders) | 3
Haemorrhoids (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 24
Odynophagia (Gastrointestinal disorders) | 2
Oesophagitis (Gastrointestinal disorders) | 2
Oral pain (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 28
Vomiting (Gastrointestinal disorders) | 13
Asthenia (General disorders) | 5
Chest pain (General disorders) | 3
Chills (General disorders) | 7
Fatigue (General disorders) | 20
Oedema (General disorders) | 3
Oedema peripheral (General disorders) | 10
Pyrexia (General disorders) | 13
Bacterial infection (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 2
Candidiasis (Infections and infestations) | 2
Clostridial infection (Infections and infestations) | 2
Device related infection (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 4
Sepsis (Infections and infestations) | 2
Contusion (Injury, poisoning and procedural complications) | 2
Excoriation (Injury, poisoning and procedural complications) | 2
Skin laceration (Injury, poisoning and procedural complications) | 3
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 4
Blood calcium decreased (Investigations) | 2
Blood creatinine increased (Investigations) | 4
Blood glucose increased (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 3
Blood potassium decreased (Investigations) | 2
International normalised ratio increased (Investigations) | 2
Neutrophil count decreased (Investigations) | 2
Weight decreased (Investigations) | 8
White blood cell count decreased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 17
Dehydration (Metabolism and nutrition disorders) | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 6
Hyperphosphataemia (Metabolism and nutrition disorders) | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 15
Hypomagnesaemia (Metabolism and nutrition disorders) | 6
Hyponatraemia (Metabolism and nutrition disorders) | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 6
Malnutrition (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 9
Dysgeusia (Nervous system disorders) | 9
Headache (Nervous system disorders) | 9
Memory impairment (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 6
Peripheral sensory neuropathy (Nervous system disorders) | 2
Sinus headache (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 5
Confusional state (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 3
Hallucination (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 7
Dysuria (Renal and urinary disorders) | 4
Haematuria (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 3
Renal failure acute (Renal and urinary disorders) | 3
Urinary retention (Renal and urinary disorders) | 2
Scrotal erythema (Reproductive system and breast disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 6
Dermatitis (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 6
Erythema (Skin and subcutaneous tissue disorders) | 4
Petechiae (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 8
Skin disorder (Skin and subcutaneous tissue disorders) | 3
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 6
Flushing (Vascular disorders) | 4
Hypertension (Vascular disorders) | 4
Hypotension (Vascular disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No